CLINICAL TRIAL: NCT05006703
Title: Breathing Retraining for Asthma Trial of Home Exercises for Teenagers (Breathe4T); Re-purposing, Refining and Feasibility - Stage 3
Brief Title: Breathing Retraining for Asthma Trial of Home Exercises for Teenagers
Acronym: Breathe4T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University of Bath (Other); Aston University (Other); University Hospital Southampton NHS Foundation Trust (Other); Asthma UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHI1071; PB-PG-0817-20038 (Other Grant/Funding Number: NIHR RfPB)
Record Dates: First submitted 2021-06-23; First posted 2021-08-16 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Adolescent Behavior; Asthma
MeSH Terms: conditions — Adolescent Behavior; Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Access to digital intervention
  Interventions: Behavioral: Breathe for Teens (Breathe4T)
- Control group (No Intervention): Usual care group

INTERVENTIONS:
Behavioral: Breathe for Teens (Breathe4T) — A digital, self-management intervention for adolescents to control their asthma using breathing retraining. The mobile-friendly website provides information about asthma, how it affects the lungs, and how breathing patterns can be dysfunctional. Information is presented using short (30sec-2min) video clips featuring physiotherapists, researchers and adolescent role models. Users are given tips about their practice, including choosing a suitable time and place and building up gradually. Users can plan and log their practice and record their confidence in using the breathing techniques. There are 8 sessions including peer-led videos demonstrating breathing exercises with voiceovers and step-by-step instructions. All features and sessions can be accessed via a main dashboard where users can tailor the intervention to allow parental involvement, reminders and a preferred format for notifications (email/text). Other features include frequently asked questions (FAQs) and a progress chart.
  Arms: Intervention group

SUMMARY:
This trial will address the impaired quality of life of young people with asthma, despite appropriate medicines. Research shows that young people report needing to calm themselves down during an asthma attack to control their breathing. Although physiotherapist- delivered breathing retraining programmes now have a clear evidence base in adults with asthma, improving quality of life, there is a lack of evidence assessing its use in younger patients. The investigators have redesigned an adult training package to make it appropriate for young people and will now assess how effective such an intervention would be in this population. This study will include young people (12-17 years) with physician diagnosed asthma. The repurposing, optimisation and acceptability of the intervention in the adolescent age group has been undertaken in Stages 1 and 2 of the Breathe 4 Teens (BREATHE4T) project. A self-guided, breathing retraining digital intervention has been developed, delivered via a mobile friendly, online platform.

The current study is a randomised, controlled feasibility trial and will provide the necessary information for a substantive cost-effectiveness trial. Participants with access to the intervention will be compared to a usual care group. Asthma and quality of life of both groups will also be assessed at baseline, 2-month and 6-month time points. At the end of the 6 months, the control group will also be given access to the website.

The online nature of this study allows recruitment from across the United Kingdom. Recruitment methods would include primary care, hospital clinics, social media and posters. AsthmaUK will also provide publicity to assist recruitment.

DETAILED DESCRIPTION:
The trial will aim to assess the acceptability, uptake and success in collecting follow up data and variance in asthma-related outcome measures. A parallel group design will be used with participants being randomised to intervention or normal management. The intervention will be a self-guided, breathing retraining digital intervention, delivered via a mobile-friendly, online platform. The intervention will continue to be used for 6 months after which both groups will be reassessed. The usual management control group will then have access to the intervention (delayed access).

ELIGIBILITY:
Inclusion Criteria:

* Young people aged 12-17 years
* Physician diagnosed asthma
* Impaired quality of life (<85)
* Under the care of a general practitioner, community or hospital practitioner for their asthma

Exclusion Criteria:

* Co-existent respiratory conditions such as bronchiectasis
* Already using breathing techniques
* Already enrolled in another interventional study
* Lack of informed consent
* Learning difficulties
* Previously involved with Stages 1 and 2 of the study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Roberts, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study webpage — https://www.southampton.ac.uk/breathe4t

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Access to digital intervention
  Breathe for Teens (Breathe4T): A digital, self-management intervention for adolescents to control their asthma using breathing retraining. The mobile-friendly website provides information about asthma and how it affects the lungs, as well as how breathing patterns can be dysfunctional. Information is presented using short (30sec-2min) video clips featuring physiotherapists, researchers and adolescent role models. Users are given tips about their practice, including choosing a suitable time and place and building up gradually. Users can plan their practice, log how their practice went and record their confidence in using the breathing techniques. There are 8 sessions including peer-led videos demonstrating breathing exercises with voice overs and step-by-step instructions. All features and sessions can be accessed via a main dashboard where users can tailor the intervention to allow parental involvement, reminders and a preferred format for notifications (email/text). Other features include frequently asked questions (FAQs) and a progress chart.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 32 | 32
Completed | 18 | 27
Not Completed | 14 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Access to digital intervention
  Breathe4T: A digital, self-management intervention for adolescents to control their asthma using breathing retraining. The mobile-friendly website provides information about asthma and how it affects the lungs, as well as how breathing patterns can be dysfunctional. Information is presented using short (30sec-2min) video clips featuring physiotherapists, researchers and adolescent role models. Users are given tips about their practice, including choosing a suitable time and place and building up gradually. Users can plan their practice, log how their practice went and record their confidence in using the breathing techniques. There are 8 sessions including peer-led videos demonstrating breathing exercises with voiceovers and step-by-step instructions. All features and sessions can be accessed via a main dashboard where users can tailor the intervention to allow parental involvement, reminders and a preferred format for notifications (email/text). Other features include FAQs and a progress chart.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Customized [Count of Participants; unit: Participants]
  Age (years): 12-14 | 13 | 16 | 29
  Age (years): 15-17 | 19 | 16 | 35
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 8 | 12 | 20
  Gender: Female | 23 | 18 | 41
  Gender: Prefer not to say / unknown | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White/English/Scottish/Welsh | 29 | 30 | 59
  Ethnicity: White other | 1 | 1 | 2
  Ethnicity: Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 32 | 32 | 64
Attended accident and emergency (A&E) in past year [Count of Participants; unit: Participants]
  No | 27 | 28 | 55
  Yes | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Asthma-specific Quality of Life
Description: PedsQL (paediatric quality of life inventory) - asthma module - presented as a total score with a higher score indicating lower problems, and therefore better quality of life. Min 0 - Max 100. Scale scores are computed as the sum of the items over the number of items answered.
Time Frame: 6 months
Population: Number analysed at 6 months is less than baseline due to loss at follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 32
score on a scale
  Baseline | 65.4 (13.2) | 65.1 (15.6)
  6 months: number analyzed (Participants) | 18 | 27
  6 months | 66.7 (11.3) | 67.4 (18.1)

2. Primary Outcome: Asthma Control
Description: Asthma control test (ACT) - presented as a total score with a lower score indicating poor control. Overall score above 19 would indicate well-controlled asthma. Min value 0 - Max 25.
Time Frame: 6 months
Population: Number analysed is different between baseline and 6 months due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 32
score on a scale
  Baseline | 17.2 (5.2) | 17.4 (4.5)
  6 months: number analyzed (Participants) | 18 | 22
  6 months | 16.9 (4.1) | 17.8 (5.2)

3. Primary Outcome: Episodes of Prescriptions of 3 or More Days of Prednisolone (or Similar)
Description: Self-reported in a healthcare utilisation questionnaire.
Time Frame: 6 months
Population: number analysed at 6 months is less than baseline due to loss to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 32
Participants
  Baseline: Yes | 9 | 11
  Baseline: No | 23 | 21
  6 months: number analyzed (Participants) | 18 | 22
  6 months: Yes | 5 | 6
  6 months: No | 13 | 16

4. Secondary Outcome: Attendance at Emergency Department for an Exacerbation of Asthma
Description: Self-reported in a healthcare utilisation questionnaire
Time Frame: 6 months
Population: Number analysed differs from baseline to 6 months due to loss to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 32
Participants
  Baseline: yes | 5 | 4
  Baseline: no | 27 | 28
  6 months: number analyzed (Participants) | 18 | 22
  6 months: yes | 0 | 2
  6 months: no | 18 | 20

5. Secondary Outcome: Hospital Admission for an Exacerbation of Asthma
Description: Self-reported in a healthcare utilisation questionnaire
Time Frame: 6 months
Population: Number analysed differs due to loss to follow-up at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 32
Participants
  Baseline: yes | 14 | 17
  Baseline: no | 18 | 15
  6 months: number analyzed (Participants) | 18 | 22
  6 months: yes | 0 | 2
  6 months: no | 18 | 20

6. Secondary Outcome: Paediatric Quality of Life
Description: Paediatric asthma quality life questionnaire (PAQLQ) - presented as a total score. Higher scores represent a better quality of life. Min value 1 - max 7.
Time Frame: 6 months
Population: Number analysed at 6 months in less than baseline due to loss at follow-up. Key finding of feasibility trial that burden of this additional paper questionnaire was not feasible.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 32 | 32
score on a scale
  Baseline | 4.5 (1.6) | 5.1 (1.5)
  6 months: number analyzed (Participants) | 6 | 12
  6 months | 5.7 (0.7) | 4.6 (1.5)

ADVERSE EVENTS:
Time Frame: 6 month trial period
Description: Adverse events are reported for both the intervention and control group during the 6 month trial period.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT05006703/Prot_SAP_000.pdf